CLINICAL TRIAL: NCT05758077
Title: A Multi-Center, Randomized, Controlled, Pivotal Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device in Patients With Acute Kidney Injury Requiring Continuous Kidney Replacement Therapy
Brief Title: Neutrophil and Monocyte Deactivation Via the SeLective CytopheretIc Device - A Randomized Clinical Trial in Acute Kidney Injury
Acronym: NEUTRALIZE-AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SeaStar Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCD-006
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
Keywords: continuous kidney replacement therapy; continuous renal replacement therapy; acute kidney injury; organ failure; inflammation; dialysis; acute tubular necrosis
MeSH Terms: conditions — Acute Kidney Injury; Inflammation; Kidney Cortex Necrosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- SCD + CKRT Arm (Experimental): In addition to standard of care CKRT therapy for these subjects, these subjects will have up to ten sequential 24-hour treatments with the Selective Cytopheretic Device (SCD) in-line with their existing CKRT circuit.
  Interventions: Device: Selective Cytopheretic Device
- CKRT Alone Arm (standard of care) (Other): This arm will receive standard of care CKRT therapy for their condition as appropriate.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Selective Cytopheretic Device — The Selective Cytopheretic Device (SCD) is comprised of tubing, connectors, and a synthetic hollow fiber membrane cartridge. The device is connected in series to a commercially available CKRT hemofilter. Blood from the CKRT circuit is diverted after the CKRT hemofilter through to the extracapillary space (ECS) of the SCD cartridge. Blood circulates through the SCD ECS and then it is returned to the patient via the venous return line of the CKRT circuit. Regional citrate anticoagulation is used for the entire CKRT and SCD blood circuit.
  The SCD cartridge incorporates a synthetic hollow fiber membrane with the ability to bind activated leukocytes to its extracapillary surface; and when used in a CKRT extracorporeal circuit in the presence of regional citrate anticoagulation, the SCD modulates inflammation.
  Other Names: SCD
  Arms: SCD + CKRT Arm
Other: Standard of Care — Standard of care CKRT for the subject's condition, as appropriate
  Arms: CKRT Alone Arm (standard of care)

SUMMARY:
This randomized, controlled, pivotal study is intended to determine whether up to ten sequential 24-hour treatments with the Selective Cytopheretic Device (SCD) will improve survival in patients with Acute Kidney Injury (AKI) requiring continuous kidney replacement therapy (CKRT) when compared to CKRT alone (standard of care). This study is further intended to determine whether SCD therapy will reduce the duration of maintenance dialysis secondary to AKI. This study will enroll approximately 200 subjects across 30 US sites. Participants will be patients in an intensive care unit (ICU) setting with a diagnosis of AKI requiring CKRT.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an ICU requiring CKRT:

  1. Must have AKI stage 2 or greater at the time of CKRT initiation.
  2. Must have been on CKRT for at least 12 hours but no greater than 48 hours at the time of enrollment.
* At least 18 years of age but not older than 80 at the time of enrollment.
* One additional life-threatening organ dysfunction present.
* Acceptable vascular access for CKRT to include adequate lumen size and length of catheters.
* Initial (non-binding) commitment to maintaining current level of care for at least 96 hours.
* C-Reactive Protein >3.5 mg/dl.

Exclusion Criteria:

* Not expected to survive next 24 hours.
* Anticipated transition to comfort measures or hospice in next 4 days.
* Terminal condition whereby the patient is not expected to survive 28 days or any condition in which therapy is regarded as futile by the PI.
* Advanced malignancy which is actively being treated or may be treated with palliative chemotherapy or radiation.
* ICU hospitalization > 14 days during this hospital admission (to include days spent at ICU of an outside hospital) at the time of screening.
* Active COVID-19 infection with a primary admission diagnosis of COVID-19.
* Chronic use of ventricular assist devices.
* ESRD requiring chronic kidney replacement therapy.
* History of CKD (greater than Stage 3).
* AKI stage 0 or stage 1 at the time of CKRT initiation.
* Non-ATN AKI diagnosis. We intend on relying on local nephrology subspecialty expertise to reasonably exclude non-ATN diagnoses based on clinical suspicions combined with prespecified objective criteria. If there is a reasonable suspicion that the subject has non-ATN AKI based on this, they will be excluded from the trial.
* Acute coronary syndromes, acute stroke, or acute major vascular compromise requiring medical or surgical interventions within 48 hours of randomization.
* Active hemorrhage requiring blood transfusions at the time of screening.
* Acute on Chronic Liver Failure.
* Suspicion of hepato-renal syndrome.
* Presence of any solid organ transplant at any time prior to admission.
* Severe burns with a modified Baux score > 100 (%TBSA+Age+17 for Inhalation Injury).
* Bone marrow transplant within the last year.
* Chronic immunosuppression with an average of >20 mg/day of prednisone or other steroid sparing immunosuppressants for the past 30 days prior to hospital admission.
* Individuals who have a history of primary or secondary immune disorders including, but not limited to, HIV or AIDS.
* Dry weight of >150kg.
* Platelet count <15,000/mm3.
* Patient is a prisoner or member of a vulnerable population.
* Patient is pregnant or breast feeding.
* Concurrent enrollment in another interventional clinical trial for an investigational drug or device.
* Need for plasmapheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of mortality or dialysis dependency at 90 days | 90 days
  The composite of death or requiring kidney replacement therapy at 90 days post randomization

SECONDARY OUTCOMES:
MAKE90 | 90 days
  Major adverse kidney events at day 90 is a composite of death, need for KRT, or persistent renal dysfunction (final serum creatinine concentration, ≥200% of the baseline value) at the 90 day follow up period
Dialysis dependence | 1 year
  Need for any form of kidney replacement therapy at one year
ICU free days in the first 28 days | 28 days
  The number of days alive and requiring ICU level of care in the 28 days after randomization for at least 24 hours
Mortality at 28 days | 28 days
  Death by day 28 post randomization

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - University of Alabama Birmingham Hospital, Birmingham, Alabama
  - Central Arkansas Veterans Healthcare, Little Rock, Arkansas
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Hospital Anschutz Medical Campus, Aurora, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - JMS Burn Center, Augusta, Georgia
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kentucky HealthCare, Lexington, Kentucky
  - Ochsner LSU Health Academic Medical Center, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - UNLV Health, Las Vegas, Nevada
  - Unversity of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Samaritan Health, Corvallis, Oregon
  - St Luke's University Hospital, Bethlehem, Pennsylvania
  - Saint Mary Medical Center, Langhorne, Pennsylvania
  - Nazareth Hospital, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - United States Army Institute of Surgical Research, JBSA Fort Sam Houston, Texas
  - Methodist Hospital Metropolitan, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Texas Health San Antonio, San Antonio, Texas
  - Sentara Health, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjellstrand CM, Gornick C, Davin T. Recovery from acute renal failure. Clin Exp Dial Apheresis. 1981;5(1-2):143-61. doi: 10.3109/08860228109076011. PMID 7333033
- [Background] Hall JW, Johnson WJ, Maher FT, Hunt JC. Immediate and long-term prognosis in acute renal failure. Ann Intern Med. 1970 Oct;73(4):515-21. doi: 10.7326/0003-4819-73-4-515. No abstract available. PMID 5506002
- [Background] VA/NIH Acute Renal Failure Trial Network; Palevsky PM, Zhang JH, O'Connor TZ, Chertow GM, Crowley ST, Choudhury D, Finkel K, Kellum JA, Paganini E, Schein RM, Smith MW, Swanson KM, Thompson BT, Vijayan A, Watnick S, Star RA, Peduzzi P. Intensity of renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Jul 3;359(1):7-20. doi: 10.1056/NEJMoa0802639. Epub 2008 May 20. PMID 18492867
- [Background] Palevsky PM, O'Connor TZ, Chertow GM, Crowley ST, Zhang JH, Kellum JA; US Department of Veterans Affairs/National Institutes of Health Acute Renal Failure Trial Network. Intensity of renal replacement therapy in acute kidney injury: perspective from within the Acute Renal Failure Trial Network Study. Crit Care. 2009;13(4):310. doi: 10.1186/cc7901. Epub 2009 Aug 11. PMID 19678919
- [Background] Van Den Noortgate N, Mouton V, Lamot C, Van Nooten G, Dhondt A, Vanholder R, Afschrift M, Lameire N. Outcome in a post-cardiac surgery population with acute renal failure requiring dialysis: does age make a difference? Nephrol Dial Transplant. 2003 Apr;18(4):732-6. doi: 10.1093/ndt/gfg043. PMID 12637642
- [Background] Liano F, Junco E, Pascual J, Madero R, Verde E. The spectrum of acute renal failure in the intensive care unit compared with that seen in other settings. The Madrid Acute Renal Failure Study Group. Kidney Int Suppl. 1998 May;66:S16-24. PMID 9580541
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Metnitz PG, Krenn CG, Steltzer H, Lang T, Ploder J, Lenz K, Le Gall JR, Druml W. Effect of acute renal failure requiring renal replacement therapy on outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2051-8. doi: 10.1097/00003246-200209000-00016. PMID 12352040
- [Background] McCarthy JT. Prognosis of patients with acute renal failure in the intensive-care unit: a tale of two eras. Mayo Clin Proc. 1996 Feb;71(2):117-26. doi: 10.4065/71.2.117. PMID 8577185
- [Background] Star RA. Treatment of acute renal failure. Kidney Int. 1998 Dec;54(6):1817-31. doi: 10.1046/j.1523-1755.1998.00210.x. PMID 9853246
- [Background] Simmons EM, Himmelfarb J, Sezer MT, Chertow GM, Mehta RL, Paganini EP, Soroko S, Freedman S, Becker K, Spratt D, Shyr Y, Ikizler TA; PICARD Study Group. Plasma cytokine levels predict mortality in patients with acute renal failure. Kidney Int. 2004 Apr;65(4):1357-65. doi: 10.1111/j.1523-1755.2004.00512.x. PMID 15086475
- [Background] Mutunga M, Fulton B, Bullock R, Batchelor A, Gascoigne A, Gillespie JI, Baudouin SV. Circulating endothelial cells in patients with septic shock. Am J Respir Crit Care Med. 2001 Jan;163(1):195-200. doi: 10.1164/ajrccm.163.1.9912036. PMID 11208646
- [Background] Himmelfarb J, McMonagle E, Freedman S, Klenzak J, McMenamin E, Le P, Pupim LB, Ikizler TA, The PICARD Group. Oxidative stress is increased in critically ill patients with acute renal failure. J Am Soc Nephrol. 2004 Sep;15(9):2449-56. doi: 10.1097/01.ASN.0000138232.68452.3B. PMID 15339994
- [Background] Camon AM, Alonso R, Munoz FJ, Cardozo C, Bernal-Maurandi J, Albiach L, Aguero D, Marcos MA, Ambrosioni J, Bodro M, Chumbita M, De la Mora L, Garcia-Pouton N, Duenas G, Hernandez-Meneses M, Inciarte A, Cuesta G, Meira F, Morata L, Puerta-Alcalde P, Rico V, Herrera S, Tuset M, Castro P, Prieto-Gonzalez S, Almuedo A, Munoz J, Mensa J, Sanjuan G, Nicolas JM, Del Rio A, Vila J, Garcia F, Martinez JA, Garcia-Vidal C, Soriano A; Hospital Clinic of Barcelona COVID-19 Research Group. C-reactive protein cut-off for early tocilizumab and dexamethasone prescription in hospitalized patients with COVID-19. Sci Rep. 2022 Mar 28;12(1):5250. doi: 10.1038/s41598-022-08882-x. PMID 35347166
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Background] Carson JL, Guyatt G, Heddle NM, Grossman BJ, Cohn CS, Fung MK, Gernsheimer T, Holcomb JB, Kaplan LJ, Katz LM, Peterson N, Ramsey G, Rao SV, Roback JD, Shander A, Tobian AA. Clinical Practice Guidelines From the AABB: Red Blood Cell Transfusion Thresholds and Storage. JAMA. 2016 Nov 15;316(19):2025-2035. doi: 10.1001/jama.2016.9185. PMID 27732721
- [Background] Compher C, Bingham AL, McCall M, Patel J, Rice TW, Braunschweig C, McKeever L. Guidelines for the provision of nutrition support therapy in the adult critically ill patient: The American Society for Parenteral and Enteral Nutrition. JPEN J Parenter Enteral Nutr. 2022 Jan;46(1):12-41. doi: 10.1002/jpen.2267. Epub 2022 Jan 3. PMID 34784064
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Nanchal R, Subramanian R, Karvellas CJ, Hollenberg SM, Peppard WJ, Singbartl K, Truwit J, Al-Khafaji AH, Killian AJ, Alquraini M, Alshammari K, Alshamsi F, Belley-Cote E, Cartin-Ceba R, Dionne JC, Galusca DM, Huang DT, Hyzy RC, Junek M, Kandiah P, Kumar G, Morgan RL, Morris PE, Olson JC, Sieracki R, Steadman R, Taylor B, Alhazzani W. Guidelines for the Management of Adult Acute and Acute-on-Chronic Liver Failure in the ICU: Cardiovascular, Endocrine, Hematologic, Pulmonary, and Renal Considerations. Crit Care Med. 2020 Mar;48(3):e173-e191. doi: 10.1097/CCM.0000000000004192. PMID 32058387
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Chung KK, Stewart IJ, Gisler C, Simmons JW, Aden JK, Tilley MA, Cotant CL, White CE, Wolf SE, Renz EM. The Acute Kidney Injury Network (AKIN) criteria applied in burns. J Burn Care Res. 2012 Jul-Aug;33(4):483-90. doi: 10.1097/BCR.0b013e31825aea8d. PMID 22688091
- [Background] Yap E, Prysyazhnyuk Y, Ouyang J, Puri I, Boutin-Foster C, Salifu M. The Implication of Dropping Race from the MDRD Equation to Estimate GFR in an African American-Only Cohort. Int J Nephrol. 2021 Nov 16;2021:1880499. doi: 10.1155/2021/1880499. eCollection 2021. PMID 34824870
- [Background] Self WH, Semler MW, Wanderer JP, Wang L, Byrne DW, Collins SP, Slovis CM, Lindsell CJ, Ehrenfeld JM, Siew ED, Shaw AD, Bernard GR, Rice TW; SALT-ED Investigators. Balanced Crystalloids versus Saline in Noncritically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):819-828. doi: 10.1056/NEJMoa1711586. Epub 2018 Feb 27. PMID 29485926
- [Background] Tumlin J, Wali R, Williams W, Murray P, Tolwani AJ, Vinnikova AK, Szerlip HM, Ye J, Paganini EP, Dworkin L, Finkel KW, Kraus MA, Humes HD. Efficacy and safety of renal tubule cell therapy for acute renal failure. J Am Soc Nephrol. 2008 May;19(5):1034-40. doi: 10.1681/ASN.2007080895. Epub 2008 Feb 13. PMID 18272842
- [Background] Ding F, Yevzlin AS, Xu ZY, Zhou Y, Xie QH, Liu JF, Zheng Y, DaSilva JR, Humes HD. The effects of a novel therapeutic device on acute kidney injury outcomes in the intensive care unit: a pilot study. ASAIO J. 2011 Sep-Oct;57(5):426-32. doi: 10.1097/MAT.0b013e31820a1494. PMID 21317636
- [Background] Tumlin JA, Galphin CM, Tolwani AJ, Chan MR, Vijayan A, Finkel K, Szamosfalvi B, Dev D, DaSilva JR, Astor BC, Yevzlin AS, Humes HD; SCD Investigator Group. A Multi-Center, Randomized, Controlled, Pivotal Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device in Patients with Acute Kidney Injury. PLoS One. 2015 Aug 5;10(8):e0132482. doi: 10.1371/journal.pone.0132482. eCollection 2015. PMID 26244978
- [Background] Tumlin JA, Chawla L, Tolwani AJ, Mehta R, Dillon J, Finkel KW, DaSilva JR, Astor BC, Yevzlin AS, Humes HD. The effect of the selective cytopheretic device on acute kidney injury outcomes in the intensive care unit: a multicenter pilot study. Semin Dial. 2013 Sep-Oct;26(5):616-23. doi: 10.1111/sdi.12032. Epub 2012 Oct 29. PMID 23106607
- [Background] Goldstein SL, Askenazi DJ, Basu RK, Selewski DT, Paden ML, Krallman KA, Kirby CL, Mottes TA, Terrell T, Humes HD. Use of the Selective Cytopheretic Device in Critically Ill Children. Kidney Int Rep. 2020 Dec 19;6(3):775-784. doi: 10.1016/j.ekir.2020.12.010. eCollection 2021 Mar. PMID 33732992
- [Background] Yessayan LT, Neyra JA, Westover AJ, Szamosfalvi B, Humes HD. Extracorporeal Immunomodulation Treatment and Clinical Outcomes in ICU COVID-19 Patients. Crit Care Explor. 2022 May 19;4(5):e0694. doi: 10.1097/CCE.0000000000000694. eCollection 2022 May. PMID 35620768
- [Background] Yessayan L, Szamosfalvi B, Napolitano L, Singer B, Kurabayashi K, Song Y, Westover A, Humes HD. Treatment of Cytokine Storm in COVID-19 Patients With Immunomodulatory Therapy. ASAIO J. 2020 Nov/Dec;66(10):1079-1083. doi: 10.1097/MAT.0000000000001239. PMID 33136592
- See also: CKD stages — https://www.davita.com/education/kidney-disease/stages
- See also: ICU Liberation Bundle — https://www.sccm.org/Clinical-Resources/ICULiberation-Home/ABCDEF-Bundles